CLINICAL TRIAL: NCT03904615
Title: A Phase I Randomized Clinical Trial of In-hospital and Post-hospital Whey Protein vs. Low Quality Protein vs. Isocaloric Placebo Supplementation to Improve Recovery From Hospitalization in Older Adults
Brief Title: Geriatric Recovery Using Inpatient and Post-hospitalization Supplementation
Acronym: GRIPS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 18-0247
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Aging
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Intervention Model Description: Parallel randomized double blind phase 1 trial of 3 interventions
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whey Protein (Active Comparator): 30 g of whey protein twice daily during hospitalization and for 30 days after discharge
  Interventions: Dietary Supplement: Whey Protein
- Collagen Protein (Active Comparator): 30 g of collagen protein twice daily during hospitalization and for 30 days after discharge
  Interventions: Dietary Supplement: Collagen Protein
- Placebo (Placebo Comparator): 30 g of maltodextrin twice daily during hospitalization and for 30 days after discharge
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Whey Protein — 30 g of whey protein in flavored water, twice daily, during hospitalization and for 30 days post-discharge
  Arms: Whey Protein
Dietary Supplement: Collagen Protein — 30 g of collagen protein in flavored water, twice daily, during hospitalization and for 30 days post-discharge
  Arms: Collagen Protein
Dietary Supplement: Placebo — 30 g of maltodextrin in flavored water, twice daily, during hospitalization and for 30 days post-discharge
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the feasibility of nutritional interventions designed to help older patients maintain physical function after being in the hospital. We will test the feasibility and effect of nutritional interventions with whey protein, collagen or placebo on functional recovery from hospitalization in community dwelling older adults.

DETAILED DESCRIPTION:
We will compare in a randomized parallel design double blind pilot phase I study the feasibility of whey protein vs. collagen vs. isocaloric placebo supplementation in older adults during an acute hospitalization for a medical condition, and the treatments' effect size on physical function after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older.
* Admitted to UTMB hospital for any acute medical condition
* English speaking

Exclusion Criteria:

* Inability to consent
* Bed or wheelchair bound prior to hospitalization
* Estimated creatinine clearance 20 ml/min or less, or end stage renal disease not on dialysis
* AST/ALT 2.5 times above the normal limit
* Active cancer
* Palliative care/Hospice
* Estimated protein intake >1.2 g/kg/day during the previous 24 hours
* Any other condition or event considered exclusionary by the PI and faculty physician

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Physical Function | Change from baseline to 30 days after discharge
  Short Physical Performance Battery (SPPB) scale, 0-12 points. 0=disabled; 12=high performance

CONTACTS AND LOCATIONS:
Overall Officials: Elena Volpi, MD, PhD, Principal Investigator — UTMB
Locations (2):
- United States (2):
  - UTMB Acute Care for Elders Unit, Galveston, Texas
  - Jennie Sealy Hospital, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No
No. This is a small Phase 1 feasibility pilot study. Risk of loss of confidentiality